CLINICAL TRIAL: NCT03507309
Title: National Institute for Health Research (NIHR) Cardiovascular Health Informatics Collaborative
Brief Title: NIHR CV Health Informatics Collaborative
Acronym: NHIC-CV
Status: Active, not recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other); Oxford University Hospitals NHS Trust (Other); University College London Hospitals (Other); University Hospital Southampton NHS Foundation Trust (Other); University Hospitals, Leicester (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Manchester University NHS Foundation Trust (Other Government); University Hospital Birmingham NHS Foundation Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other); Blackpool Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Jamil Mayet, Professor of Cardiology, Imperial College London
Other Study IDs: 174052; 16/HRA/3327 (Other: Integrated Research Application System)
Record Dates: First submitted 2018-02-23; First posted 2018-04-25 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-07

CONDITIONS: Troponin; Age; Mortality; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unselected cohort of patients who had a troponin measured: Patients who presented to hospital during the study period (2010-17) and had at least one troponin blood test measured.

SUMMARY:
The National Institute for Health Research (NIHR) Cardiovascular Health Informatics Collaborative is an observational, multi-centre and longitudinal study of clinical data from collaborating hospitals. A dataset of the longitudinal record for patients who presented with a suspected acute coronary syndrome, characterised by the request of a troponin test, has been developed (NHIC-Troponin Study).

DETAILED DESCRIPTION:
The NHIC Cardiovascular Project in the United Kingdom was established to enable the sharing and repurposing of routinely captured clinical data for re-use in research. Data sharing for this study has been enabled by establishing a data sharing agreement between each of the collaborating hospitals. The data sharing agreement allows data to be shared between National Health Service (NHS) hospitals in accordance with an anonymisation and de-identification profile approved by each information governance department, ensuring that patient identities are protected. Ethics approval for each dataset has been obtained which detailed the further de-identification steps to ensure that research datasets are fully anonymised.

The cardiovascular theme clinical leads developed a standard target data model specification to capture the longitudinal record for patients who presented with a suspected acute coronary syndrome, characterised by the request of a troponin test (NHIC-Troponin Study). The data model was patient centric allowing for minor discrepancies between dataset areas such as missing discharges or test results returning outside of episodes of care. The model included 156 data points, grouped into demographics, cardiovascular risk factors, emergency department attendance and inpatient episodes, biochemistry, revascularisation and mortality. All patients were followed up on the NHS Spine Application, Summary Care Record until death or censoring on 1st April 2017.

This dataset comprised all patients who had a troponin measured at each of the five major academic centres between 2010 (2008 for University College Hospital) and 2017. The investigators identified a total of 257948 patient records who underwent troponin testing during the study period.

A Committee of Experts validates the protocol methodology and supervises the data management. A Steering Committee oversees study proposals including hypotheses, study design and statistical analyses including planned outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to one of the collaborating hospitals.

Exclusion Criteria:

* Nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with electronic records at collaborating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 257948 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Mayet, Principal Investigator — Imperial College London

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual electronic patient record data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will me made available from study completion date.
Access Criteria: Data access requests will be reviewed by a Steering Committee from the participating Biomedical Research Centres. Requesters will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Scott JK, Johnson T, Caskey FJ, Bailey P, Selman LE, Mulla A, Glampson B, Davies J, Papdimitriou D, Woods K, O'Gallagher K, Williams B, Asselbergs FW, Mayer EK, Lee R, Herbert C, Grant SW, Curzen N, Squire I, Kharbanda R, Shah A, Perera D, Patel RS, Channon K, Mayet J, Kaura A, Ben-Shlomo Y. Association between kidney function, frailty and receipt of invasive management after acute coronary syndrome. Open Heart. 2024 Oct 9;11(2):e002875. doi: 10.1136/openhrt-2024-002875. PMID 39384342
- [Derived] Kaura A, Hartley A, Panoulas V, Glampson B, Shah ASV, Davies J, Mulla A, Woods K, Omigie J, Shah AD, Thursz MR, Elliott P, Hemmingway H, Williams B, Asselbergs FW, O'Sullivan M, Lord GM, Trickey A, Sterne JA, Haskard DO, Melikian N, Francis DP, Koenig W, Shah AM, Kharbanda R, Perera D, Patel RS, Channon KM, Mayet J, Khamis R. Mortality risk prediction of high-sensitivity C-reactive protein in suspected acute coronary syndrome: A cohort study. PLoS Med. 2022 Feb 22;19(2):e1003911. doi: 10.1371/journal.pmed.1003911. eCollection 2022 Feb. PMID 35192610
- [Derived] Kaura A, Panoulas V, Glampson B, Davies J, Mulla A, Woods K, Omigie J, Shah AD, Channon KM, Weber JN, Thursz MR, Elliott P, Hemingway H, Williams B, Asselbergs FW, O'Sullivan M, Kharbanda R, Lord GM, Melikian N, Patel RS, Perera D, Shah AM, Francis DP, Mayet J. Association of troponin level and age with mortality in 250 000 patients: cohort study across five UK acute care centres. BMJ. 2019 Nov 20;367:l6055. doi: 10.1136/bmj.l6055. PMID 31748235
- See also: Creating 'big data' from health records to improve care — http://www.imperial.ac.uk/news/176510/creating-aposbig-data-from-health-records/

RESULTS

PARTICIPANT FLOW:
Groups:
- Unselected Cohort of Patients Who Had a Troponin Measured: A total of 257 948 patients who presented to hospital during the study period (2010-17) and had at least one troponin blood test measured.
Period: Overall Study
Arm/Group | Unselected Cohort of Patients Who Had a Troponin Measured
Started | 257948
Completed | 257948
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Unselected Cohort of Patients Who Had a Troponin Measured
Number analyzed (Participants) | 257948
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [50 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115230
  Male | 142718
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 147321
  South Asian | 7169
  Black | 19925
  Other | 23401
  Missing | 60132
Region of Enrollment [Number; unit: participants]
  United Kingdom | 257948

OUTCOME MEASURES:

1. Primary Outcome: Mortality, All-cause
Description: Number of patients who died (from any cause) including in-hospital, short-term and long-term mortality
Time Frame: Hospital admission to 3 years follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Unselected Cohort of Patients Who Had a Troponin Measured
Number analyzed (Participants) | 257948
Participants | 55850

2. Secondary Outcome: Acute Revascularisation
Description: Acute revascularisation will be defined as having PCI or CABG in the time window between 48 hours before and 3 months after the first troponin measurement. This will account for patients who had revascularisation, in particular PCI, as an emergency prior to their first troponin blood test and to capture revascularisation, in particular CABG, performed as an outpatient following their index admission.
Time Frame: 3 months follow-up
Population: 134,517 accounts for the number of patients 'admitted' to hospital, who had a troponin measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Unselected Cohort of Patients Who Had a Troponin Measured
Number analyzed (Participants) | 134517
Participants | 17444

ADVERSE EVENTS:
Time Frame: Last refresh for troponin dataset was April 2017, reflecting 7 years of follow-up
Description: As the National Institute for Health Research Health Informatics Collaborative (NIHR HIC) involves collecting routine patient data from electronic health care records, there are no adverse events being collected in relation to a new intervention as part of a trial. The only adverse event that was routinely collected for all patients was all-cause mortality.
Arm/Group | Unselected Cohort of Patients Who Had a Troponin Measured
All-Cause Mortality (participants affected / at risk) | 55850/257948
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT03507309/Prot_SAP_000.pdf